CLINICAL TRIAL: NCT01500135
Title: A Randomized, Open Label, Parallel-group, Multi-center Trial to Compare Efficacy and Safety of TachoSil® Versus Surgicel® Original for the Secondary Hemostatic Treatment of Needle Hole Bleeding in Vascular Surgery
Brief Title: Comparison of Efficacy and Safety of TachoSil® Versus Surgicel® Original for the Secondary Hemostatic Treatment of Needle Hole Bleeding in Vascular Surgery
Acronym: VASUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TC-2402-039-SP; U1111-1163-1653 (Registry Identifier: WHO)
Record Dates: First submitted 2011-12-21; First posted 2011-12-26 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2016-12

CONDITIONS: Bleeding
Keywords: Vascular Surgery; Secondary treatment of needle hole bleeding; Subjects undergoing vascular surgery and who need supportive treatment in order to control bleeding
MeSH Terms: conditions — Hemorrhage | interventions — TachoSil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TachoSil® (Experimental): TachoSil® absorbable patches, applied topically, once, intraoperatively to stop bleeding. The patches were lightly compressed against the suture line for 3 minutes. The number of patches used was determined by the surgeon based on the size of the wound. If bleeding did not stop after 5 minutes treatment was repeated.
  Interventions: Drug: TachoSil®
- Surgicel® Original (Active Comparator): Surgicel® Original absorbable patches, applied topically, once, intraoperatively to stop bleeding. The patches were lightly compressed against the suture line for 3 minutes. The number of patches used was determined by the surgeon based on the size of the wound. If bleeding did not stop after 5 minutes treatment was repeated.
  Interventions: Drug: Surgicel® Original

INTERVENTIONS:
Drug: TachoSil® — TachoSil® is a sterile, ready-to-use, absorbable patch for intra-operative topical application. It consists of an equine collagen patch coated with fibrin glue components: human fibrinogen and human thrombin.
  Arms: TachoSil®
Drug: Surgicel® Original — Surgicel® Original is an absorbable hemostat (oxidized regenerated cellulose)
  Arms: Surgicel® Original

SUMMARY:
Present trial is the third study that in combination with two completed studies (one being a trial in hepatic resection surgery also comparing TachoSil® and Surgicel® Original) targeted toward providing clinical safety and efficacy data to support extending the current label of TachoSil® to a general hemostasis indication across several surgical procedures and organ systems in the USA.

DETAILED DESCRIPTION:
The drug being tested in this study is called TachoSil®. TachoSil® was used to treat people undergoing scheduled subacute vascular surgery. This study looked at how well TachoSil® patches stopped bleeding at the surgical site compared to Surgicel® Original patches.

The study enrolled 150 patients. Participants were randomly assigned (by chance, like flipping a coin) to one of the two open label treatment groups in a 2:1 ratio:

* TachoSil®
* Surgicel® Original

This multi-center trial was conducted in the United States. The overall time to participate in this study was approximately 6 months. Participants made multiple visits to the clinic, including safety follow-up visits at 1, 3 and 6 months after surgery.

ELIGIBILITY:
Main Inclusion Criteria:

* Planned elective and subacute procedures with a polytetrafluoroethylene (PTFE) graft including at least one expected end-to-side anastomosis of a PTFE graft to the femoral artery (e.g. femoral-femoral cross-over, aorto-(bi)femoral, axillo-(bi)femoral, femoro-popliteal, femoro-crural bypass grafting), a PTFE patch angioplasty of the femoral artery, or an end-to-side anastomosis of a PTFE graft to an upper extremity artery in connection with arteriovenous bypass grafting for dialysis access.
* The evaluation site for the planned femoral anastomosis must be a de novo site.
* The participant must be heparinized during surgery.

Intra-operatively (before randomization)

* The participant has a need for secondary hemostatic treatment
* Verification of the evaluation site being a de novo site
* Verification of the surgical procedure performed as being either an end-to-side or PTFE patch angioplasty.

Main Exclusion Criteria:

* Thrombolytic therapy administered within 12 hours before surgery (e.g. the recombinant tissue plasminogen activator (rt-PA) Alteplase).
* Liver cirrhosis.

Intra-operatively (before randomization)

* Severe bleeding at the anastomosis of the arterial bypass using PTFE graft prosthesis or the PTFE patch angioplasty
* No bleeding (dry surgical field) at the targeted application area
* Disseminated intravascular coagulopathy (DIC)
* Application of topical hemostatic material including fibrin sealant/glue on the evaluation site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-03; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (37):
- United States (37):
  - Nycomed Investigational Site, Birmingham, Alabama
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Long Beach, California
  - Nycomed Investigational Site, Los Angeles, California
  - Los Angeles, California
  - Loveland, Colorado
  - Jacksonville, Florida
  - Nycomed Investigational Site, Austell, Georgia
  - Austell, Georgia
  - Skokie, Illinois
  - Nycomed Investigational Site, Springfield, Illinois
  - Springfield, Illinois
  - Nycomed Investigational Site, Lexington, Kentucky
  - Lexington, Kentucky
  - Worcester, Massachusetts
  - Southfield, Michigan
  - St Louis, Missouri
  - Hackensack, New Jersey
  - East Setauket, New York
  - Flushing, New York
  - Nycomed Investigational Site, New York, New York
  - New York, New York
  - The Bronx, New York
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Toledo, Ohio
  - Portland, Oregon
  - Nycomed Investigational Site, Galveston, Texas
  - Galveston, Texas
  - Nycomed Investigational Site, Houston, Texas
  - Houston, Texas
  - Lubbock, Texas
  - Nycomed Investigational Site, Bellevue, Washington
  - Bellevue, Washington
  - Charleston, West Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 23 investigative sites in the United States from 09 March 2012 to 16 December 2015.
Pre-assignment Details: Participants who were elected for planned or subacute vascular surgery were enrolled in a 2:1 ratio to treatment groups: TachoSil® or Surgicel® Original.
Period: Overall Study
Arm/Group | TachoSil® | Surgicel® Original
Started | 100 | 50
Completed | 83 | 39
Not Completed | 17 | 11
Not completed — Withdrawal of Consent | 4 | 0
Not completed — Lost to Follow-up | 6 | 4
Not completed — Fatal Adverse Event (AE) | 5 | 5
Not completed — Principal Investigator (PI) Discretion | 1 | 0
Not completed — Patient Missed Scheduled Appointments | 0 | 1
Not completed — Participant was a Safety Concern | 1 | 0
Not completed — Patient Unable to Make Follow-up Visit | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | TachoSil® | Surgicel® Original | Total
Number analyzed (Participants) | 100 | 50 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (10.25) | 67.6 (12.87) | 66.5 (11.18)
Age, Customized [Number; unit: participants]
  ≤65 years | 48 | 22 | 70
  >65 years | 52 | 28 | 80
Gender [Count of Participants; unit: Participants]
  Female | 33 | 26 | 59
  Male | 67 | 24 | 91
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian | 79 | 34 | 113
  Asian | 0 | 1 | 1
  Black or African American | 21 | 10 | 31
  Other | 0 | 4 | 4
  Missing | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 4 | 6 | 10
  Non-Hispanic or Latino | 95 | 42 | 137
  Unknown | 1 | 1 | 2
  Missing | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 100 | 50 | 150
Height [Mean (Standard Deviation); unit: cm] — Population: Baseline height data is not available for 1 participant.
  cm
    number analyzed (Participants) | 99 | 50 | 149
    (all) | 171.70 (10.197) | 166.85 (10.381) | 170.07 (10.479)
Weight [Mean (Standard Deviation); unit: kg] — Population: Baseline weight data is not available for 1 participant.
  kg
    number analyzed (Participants) | 99 | 50 | 149
    (all) | 81.15 (18.738) | 76.20 (21.935) | 79.49 (19.932)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Baseline BMI data is not available for 1 participant.
  kg/m^2
    number analyzed (Participants) | 99 | 50 | 149
    (all) | 27.45 (5.702) | 27.13 (6.246) | 27.34 (5.871)
Fertility Status [Number; unit: participants]
  Menstrual | 2 | 1 | 3
  Postmenstrual | 15 | 15 | 30
  Surgically Sterile | 16 | 10 | 26
  Not Applicable | 67 | 24 | 91

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Intra-operative Hemostasis at the Evaluation Site Within 3 Minutes After Application of the Randomized Treatment
Description: After application of Investigational Medicinal Product (IMP) light pressure was applied to the IMP with e.g. gauze pads. The first assessment of hemostasis was at minute 3: the pressure was carefully relieved, and the area was observed for visual bleeding at the site of the IMP. If no bleeding was visible, hemostasis was obtained and recorded.
Time Frame: Within 3 minutes
Population: Full Analysis Set (FAS) included all randomized participants. The endpoint for one participant on TachoSil® was missing; it was assumed that hemostasis was not reached within 3 minutes.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TachoSil® | Surgicel® Original
Number analyzed (Participants) | 100 | 50
percentage of participants | 26.0 [17.7 to 35.7] | 18.0 [8.6 to 31.4]
Statistical Analysis 1: Comparison: TachoSil® vs Surgicel® Original; Test type: Superiority or Other; p = 0.276, Regression, Logistic — Logistic regression model with treatment, type of surgery (Peripheral Arterial Disease, Arterio Venous Graft) and current use of Clopidogrel or other similar anti-platelet drugs (yes/no) as covariates; Odds Ratio (OR) = 1.62, 95% CI 2-sided [0.68 to 3.88], Standard Error of Mean 0.72

2. Secondary Outcome: Percentage of Participants With Intra-operative Hemostasis at the Evaluation Site Within 5 Minutes After Application of the Randomized Treatment
Description: After application of Investigational Medicinal Product (IMP) light pressure was applied to the IMP with e.g. gauze pads. If hemostasis was not obtained at minute 3, pressure was immediately reapplied. Hemostasis was re-assessed at minutes 4 and 5.
Time Frame: Within 5 minutes
Population: FAS included all randomized participants. The endpoint for one participant on TachoSil® was missing; it was assumed that hemostasis was not reached within 5 minutes.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TachoSil® | Surgicel® Original
Number analyzed (Participants) | 100 | 50
percentage of participants | 39.0 [29.4 to 49.3] | 42.0 [28.2 to 56.8]
Statistical Analysis 1: Comparison: TachoSil® vs Surgicel® Original; Test type: Superiority or Other; p = 0.684, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.40 to 1.82], Standard Error of Mean 0.33

3. Secondary Outcome: Time to Intra-operative Hemostasis Within 10 Minutes at the Evaluation Site After Application of the Randomized Treatment
Description: After application of Investigational Medicinal Product (IMP) light pressure was applied to the IMP with e.g. gauze pads. Hemostasis was assessed at 3, 4, and 5 minutes. If hemostasis was not obtained after 5 minutes a second application of IMP was applied with 3 minutes of light pressure and hemostasis was re-assessed at 8, 9 and 10 minutes.
Time Frame: Within 10 minutes
Population: FAS included all randomized participants. Participants who did not achieve hemostasis by 10 minutes were censored.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | TachoSil® | Surgicel® Original
Number analyzed (Participants) | 100 | 50
minutes | 8.0 (18.87) [8.0 to 9.0] | 8.0 (14.63) [5.0 to 10.0]
Statistical Analysis 1: Comparison: TachoSil® vs Surgicel® Original; Test type: Superiority or Other; p = 0.684, Proportional Hazard Model — P-value was adjusted using Hochberg's adjustment for multiplicity; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.7 to 1.8], Standard Error of Mean 0.24

ADVERSE EVENTS:
Time Frame: From the signing of informed consent to the follow-up visit (Up to 6 Months)
Description: Safety Population included all randomized participants who received treatment. At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TachoSil® | Surgicel® Original
Serious Adverse Events (participants affected / at risk) | 49/99 | 19/50
Other Adverse Events (participants affected / at risk) | 52/99 | 28/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TachoSil® (N=99) | Surgicel® Original (N=50)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 4 | 3
Cardiac failure congestive (Cardiac disorders) | 3 | 1
Cardiomyopathy (Cardiac disorders) | 2 | 0 — One treatment-emergent death occurred during treatment with TachoSil® and is not related.
Angina unstable (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1 — One treatment-emergent death occurred during treatment with Surgicel® Original and is not related.
Cor pulmonale (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 — One treatment-emergent death occurred during treatment with TachoSil® is not related.
Atrial fibrillation (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal mass (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatic mass (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Impaired healing (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1 — One treatment-emergent death occurred during treatment with Surgicel® Original and is not related.
Pain (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 6 | 0
Wound infection (Infections and infestations) | 5 | 0
Sepsis (Infections and infestations) | 4 | 1 — One treatment-emergent death occurred during treatment with TachoSil® and one treatment-emergent death occurred during treatment with Surgicel® Original and are not related.
Cellulitis (Infections and infestations) | 2 | 0
Groin infection (Infections and infestations) | 2 | 0
Osteomyelitis (Infections and infestations) | 2 | 0
Abscess limb (Infections and infestations) | 1 | 0
Arteriovenous graft site infection (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Epstein-Barr virus infection (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 0 | 2
Haematoma infection (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 2
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 5 | 1
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 4 | 2
Vascular graft occlusion (Injury, poisoning and procedural complications) | 3 | 2
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Incision site complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 0
Graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — One treatment-emergent death occurred during treatment with TachoSil® is not related.
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cranial nerve paralysis (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Lacunar infarction (Nervous system disorders) | 1 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 3 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 3 — One treatment-emergent death occurred during treatment with Surgicel® Original and is not related.
Chronic kidney disease (Renal and urinary disorders) | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — One treatment-emergent death occurred during treatment with TachoSil® is not related.
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — One treatment-emergent death occurred during treatment with Surgicel® Original and is not related.
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Haematoma (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 2 | 1
Peripheral ischaemia (Vascular disorders) | 2 | 2
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Steal syndrome (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
Aortic aneurysm rupture (Vascular disorders) | 0 | 1
Dry gangrene (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 1
Reperfusion injury (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TachoSil® (N=99) | Surgicel® Original (N=50)
Anaemia (Blood and lymphatic system disorders) | 14 | 6
Atrial fibrillation (Cardiac disorders) | 5 | 0
Constipation (Gastrointestinal disorders) | 11 | 5
Nausea (Gastrointestinal disorders) | 7 | 0
Oedema peripheral (General disorders) | 10 | 0
Peripheral swelling (General disorders) | 3 | 3
Urinary tract infection (Infections and infestations) | 9 | 4
Seroma (Injury, poisoning and procedural complications) | 3 | 4
Wound dehiscence (Injury, poisoning and procedural complications) | 3 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 3
Insomnia (Psychiatric disorders) | 0 | 3
Urinary retention (Renal and urinary disorders) | 3 | 6
Hypotension (Vascular disorders) | 11 | 5
Hypertension (Vascular disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.